CLINICAL TRIAL: NCT01105325
Title: Evaluation of Compliance With Management of Acute Coronary Syndrome on Discharge From Cardiac Intensive Care (CIC) - Electronic Measurement of Compliance
Brief Title: Evaluation of Compliance With Management of Acute Coronary Syndrome on Discharge From Cardiac Intensive Care
Acronym: SCAVANCE
Status: Terminated | Type: Observational
Why Stopped: due to poor patient recruitment
Sponsor: AstraZeneca (Industry)
Responsible Party: MCMD, AstraZeneca
Other Study IDs: NIS-CFR-CRE-2010/1
Record Dates: First submitted 2010-03-25; First posted 2010-04-16 (Estimated); Last update posted 2010-10-04 (Estimated); Status verified 2010-10

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome; treatment compliance; cardiac intensive care unit; secondary prevention; cardiac intensive care unit (CIC); compliance; intensive care
MeSH Terms: conditions — Acute Coronary Syndrome; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To study compliance with secondary prevention during the first months following discharge from the cardiac intensive care unit (CIC) of patients experiencing a first episode of acute coronary syndrome : quantitative compliance over 3 months with the two principal treatments of the prescription (a statin - rosuvastatin, Crestor® and a platelet aggregation inhibitor - clopidogrel, Plavix®), using an electronic measure system ("intelligent blister" pack®);

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the CIC unit for a first episode of acute coronary syndrome, in whom the CIC cardiologist considers that Crestor® -rosuvastatin is the most appropriate statin, in combination with a platelet aggregation inhibitor (Plavix®-clopidogrel)
* Patient giving his/her oral consent to participate in the study.
* Patient not previously treated by a lipid-lowering drug.

Exclusion Criteria:

* Patient with a known history of coronary heart disease.
* Patient whose treatment on discharge comprises only one of the two study treatments
* Patient participating or who has participated in the previous 3 months in a biomedical research study in cardiology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First 10 patients admitted to the CIC unit for a first episode of acute coronary syndrome, in whom the CIC cardiologist considers that Crestor® - rosuvastatin is the most appropriate statin for management in hospital, in combination with a platelet aggregation inhibitor (Plavix® - clopidogrel).
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
To measure, using an electronic system ("intelligent blister pack®"), the duration of treatment and number of treatment intake per day over 3 months with statin and oral antiplatelet therapy following an inaugural acute coronary syndrome. | 3 months / every day

SECONDARY OUTCOMES:
Analysis of the duration of treatment and number of treatment intake per day at 1 month and 2 months with a statin and a platelet aggregation inhibitor, using an electronic system ("intelligent blister pack®"). | 1 and 2 months / every day
Describe global compliance with the entire prescription over 6 months | 6 months / Once at 6 months follow-up
Determine the factors influencing compliance with treatment on discharge from CIC (discharge treatment including a statin - rosuvastatin, Crestor® and a platelet aggregation inhibitor - clopidogrel, Plavix®). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Piedbois, Study Director — AstraZeneca
Locations (49):
- France (49):
  - Research Site, Antony
  - Research Site, Argenteuil
  - Research Site, Arras
  - Research Site, Avignon
  - Research Site, Bayonne
  - Research Site, Boulogne-Billancourt
  - Research Site, Bourges
  - Research Site, Caen
  - Research Site, Cholet
  - Research Site, Clamart
  - Research Site, Colmar
  - Research Site, Creil
  - Research Site, Dijon
  - Research Site, Eaubonne
  - Research Site, Épernay
  - Research Site, La Rochelle
  - Research Site, La Tronche
  - Research Site, Le Chesnay
  - Research Site, Le Coudray
  - Research Site, Le Plessis-Robinson
  - Research Site, Lens
  - Research Site, Libourne
  - Research Site, Lomme
  - Research Site, Lorient
  - Research Site, Lyon
  - Research Site, Mantes-la-Jolie
  - Research Site, Marseille
  - Research Site, Metz
  - Research Site, Montfermeil
  - Research Site, Neuilly-sur-Seine
  - Research Site, Nevers
  - Research Site, Niort
  - Research Site, Orléans
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Perpignan
  - Research Site, Pessac
  - Research Site, Périgueux
  - Research Site, Reims
  - Research Site, Rodez
  - Research Site, Saint-Nazaire
  - Research Site, Salouël
  - Research Site, Schiltigheim
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Troyes
  - Research Site, Valence
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Villeneuve-Saint-Georges